CLINICAL TRIAL: NCT03065231
Title: Lumbar Drainage Compared With Extraventricular Drainage of Cerebral Spinal Fluid in Treatment of Patients With Subarachnoid Hemorrhage - a Prospective Randomized Controlled Trial
Brief Title: Lumbar Drain vs Extraventricular Drain to Prevent Vasospasm in Subarachnoid Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Alexander A. Khalessi MD MS FAANS, Acting Clinical Chief of Neurosurgery, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160719
Record Dates: First submitted 2017-02-21; First posted 2017-02-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Vasospasm, Intracranial; Subarachnoid Hemorrhage
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: There will be two arms of the study: patients randomly assigned to LD and patients randomly assigned to EVD. Randomization will account for Fisher Grade. The two treatment arms will have CSF diversion for 7 days. For patients treated with lumbar drain, patients will have CSF drainage of 10cc/hour for lumbar drain while patients treated with EVD at 15cm above the tragus.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the type of intervention that took place.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EVD (Active Comparator): Patients will have extraventricular drain to manage CSF subarachnoid blood.
  Interventions: Device: Extraventricular Drain
- LD (Active Comparator): Patients will have lumbar drain to manage CSF subarachnoid blood.
  Interventions: Device: Lumbar Drain

INTERVENTIONS:
Device: Extraventricular Drain — As mentioned above, intervention will take place to promote subarachnoid blood diversion from cerebrospinal fluid after ruptured intracranial aneurysm.
  Arms: EVD
Device: Lumbar Drain
  Arms: LD

SUMMARY:
Vasospasm is a common complication after rupture of intracranial aneurysms causing devastating neurologic deficits and death. Vasospasm has been directly associated with the amount of subarachnoid blood inside the basal cisterns. Prior literature has attempted to refine treatment of ruptured intracranial aneurysms but does not have clear guidelines on the optimal method to drain subarachnoid blood. Two methods, extraventricular drain (EVD) and lumbar drain (LD) have been compared retrospectively yet remain controversial as to which method is optimal in reducing subarachnoid blood and preventing vasospasm. This study would be a prospective randomized trial in which patients would be assigned to EVD or LD and observed to see if one method of intervention is associated with preventing clinical vasospasm, decreasing subarachnoid blood, shortening overall ICU stay, and reducing the need for a permanent ventriculoperitoneal shunt. The conclusions of this study may identify an optimal treatment modality to benefit all future patients with ruptured intracranial aneurysms.

DETAILED DESCRIPTION:
This study will be a prospective randomized controlled trial. Participants will be patients admitted at UCSD Hillcrest or Thornton Hospital for subarachnoid hemorrhage. Patients will be recruited by the Endovascular Neurosurgical treatment team. Since there are no existing guidelines existing for procedural drainage of subarachnoid blood from the intracranial cisterns, patients are currently treated with either lumbar drain or extraventricular drain. This study would randomize the process of assigning patients to either LD or EVD as part of their treatment package for subarachnoid hemorrhage.

Both EVD and LD are regularly performed at UCSD. Both procedures are equally likely to take place if patients do not have randomization. There is currently no gold standard that dictates whether EVD should be done over LD and vice versa.

Patients will be consented to partake in the study while they are also consented for their usual care in SAH. Briefly, inclusion criteria are patients with Fisher Grade II, III, IV SAH or any aneurysmal SAH patients with radiographic evidence of hydrocephalus. Briefly, exclusion criteria are patients with obstructive hydrocephalus or mass lesion that would preclude lumbar drain placement. Pregnant patients or minors of age <18 will not be included in this study.

There will be two arms of the study: patients randomly assigned to LD and patients randomly assigned to EVD. Randomization will account for Fisher Grade. The two treatment arms will have CSF diversion for 7 days. For patients treated with lumbar drain, patients will have CSF drainage of 10cc/hour for lumbar drain while patients treated with EVD at 15cm above the tragus.

Both an extraventricular drain and a lumbar drain are defined as significant risk devices however both devices are FDA approved and will be utilized in the exact manner that they are intended. Both devices are already regularly utilized and a part of the standard of care for sub arachnoid hemorrhage management and will not be utilized in any novel way. LD and EVD assignment will be randomized through the protocol of the study.

Data will be collected via electronic medical record and will assess patient age, patient presenting Hess grade and clinical improvement post cerebrospinal fluid diversion, aneurysmal bleed day on presentation, method and technical success of securing aneurysm (clip versus coil), size and location of aneurysm, discharge disposition and clinical exam (NIH Stroke Scale), complications (tract hemorrhage or infection), need for intra-arterial management of vasospasm.

Expected Sample size in this study will include approximately 200 patients in which half of patients included in this study will be treated with LD and the other half treated with EVD. The number of estimated patients is calculated from the annual incidence of SAH received at UCSD hospitals. The facilities that are available for this project include UCSD Hillcrest Hospital, UCSD Thornton Hospital, and the UCSD Endovascular Neurosurgery suite.

The primary outcome of this study will be time to clearance of acute cisternal blood by surveillance CT (stratified by presenting Fischer Grade), need for endovascular treatment of vasospasm or stroke from vasospasm, time spent in the critical care unit, and need for ventriculoperitoneal shunt.

Regarding CT scans; Surveillance CTs are standard of care. They are typically performed on the day of device placement and subsequent imaging takes place pending clinical resolution of the patient. For most patients, they have an additional CT scan 1-2 days after initial device placement and a final scan on the 7th day of device placement. If clinical condition deteriorates, patients will have an additional scan to monitor for intracranial bleeding. The scans are performed for the clinical purpose of monitoring resolution of intracranial injury. This study would collect the data obtained from the scans.

The total exposure resulting from these imaging studies is calculated to be approximately 10 mSv. Additional head CT may be performed if clinically indicated with exposure 2.5 mSv per scan. Fluoroscopy is not routinely used, however if clinically indicated, may be utilized during lumbar drainage procedure with radiation exposure 1.5 mSv per minute. This amount is more than one would receive from one year of natural exposure in the San Diego area, which is approximately 1.6 mSv. Cumulative exposure from radiation may increase a person's risk of developing certain types of cancer in the future. This imaging is determined to be part of routine care and management of SAH. In this study, we will be merely collecting data from these images to determine clinical incidence of vasospasm and resolution of cisternal bleeding.

DSM criteria were derived from Al Tamimi et al. The initial power calculation was based off of the Al Tamimi et at study 9 that demonstrated that for 85% power, 105 patients were required in each arm of the trial. Interim analysis will be performed after recruiting 40 patients in order to establish adverse effects and an additional reevaluation at 100 patients to determine if one arm of the study is superior to the other. If this is identified, the trial will be stopped at recruitment of 100 patients. Statistical analysis will continue throughout the trial. If statistically significant differences between both arms of the study are identified earlier in the enrollment process, the study will be discontinued. Monitoring will take place internally in which the differences between the two groups will be examined for each additional 5 patients added to both groups. Internal monitoring will take place by (D.R.S.D., A.W., R.R., A.K., S.P.)

Statistical methods to evaluate data include chi square test, using independent t tests for normal numerical data, and comparing categorical data with Fisher exact test. P value of .05 will be considered clinically significant in this study.

ELIGIBILITY:
Inclusion Criteria:

* patients received at the UCSD Medical Center with grade II, III, IV subarachnoid hemorrhage or patients with aneurysmal SAH with radiographic evidence.

Exclusion Criteria:

* patients under the age of 18, excluding minors from this study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2027-01-04 (Estimated); Study Completion 2027-01-04 (Estimated)

PRIMARY OUTCOMES:
Vasopasm | 0-14 days
  Clinical and Radiographic incidence of vasospasm after ruptured intracranial aneurysm

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charpentier C, Audibert G, Guillemin F, Civit T, Ducrocq X, Bracard S, Hepner H, Picard L, Laxenaire MC. Multivariate analysis of predictors of cerebral vasospasm occurrence after aneurysmal subarachnoid hemorrhage. Stroke. 1999 Jul;30(7):1402-8. doi: 10.1161/01.str.30.7.1402. PMID 10390314
- [Background] Kassell NF, Sasaki T, Colohan AR, Nazar G. Cerebral vasospasm following aneurysmal subarachnoid hemorrhage. Stroke. 1985 Jul-Aug;16(4):562-72. doi: 10.1161/01.str.16.4.562. PMID 3895589
- [Background] Pluta RM, Hansen-Schwartz J, Dreier J, Vajkoczy P, Macdonald RL, Nishizawa S, Kasuya H, Wellman G, Keller E, Zauner A, Dorsch N, Clark J, Ono S, Kiris T, Leroux P, Zhang JH. Cerebral vasospasm following subarachnoid hemorrhage: time for a new world of thought. Neurol Res. 2009 Mar;31(2):151-8. doi: 10.1179/174313209X393564. PMID 19298755
- [Background] Shishido T, Suzuki R, Qian L, Hirakawa K. The role of superoxide anions in the pathogenesis of cerebral vasospasm. Stroke. 1994 Apr;25(4):864-8. doi: 10.1161/01.str.25.4.864. PMID 8160234
- [Background] Reilly C, Amidei C, Tolentino J, Jahromi BS, Macdonald RL. Clot volume and clearance rate as independent predictors of vasospasm after aneurysmal subarachnoid hemorrhage. J Neurosurg. 2004 Aug;101(2):255-61. doi: 10.3171/jns.2004.101.2.0255. PMID 15309916
- [Background] Friedman JA, Goerss SJ, Meyer FB, Piepgras DG, Pichelmann MA, McIver JI, Toussaint LG 3rd, McClelland RL, Nichols DA, Atkinson JL, Wijdicks EF. Volumetric quantification of Fisher Grade 3 aneurysmal subarachnoid hemorrhage: a novel method to predict symptomatic vasospasm on admission computerized tomography scans. J Neurosurg. 2002 Aug;97(2):401-7. doi: 10.3171/jns.2002.97.2.0401. PMID 12186469
- [Background] Maeda Y, Shirao S, Yoneda H, Ishihara H, Shinoyama M, Oka F, Sadahiro H, Ueda K, Sano Y, Kudomi S, Hayashi Y, Shigeeda T, Nakano K, Koizumi H, Nomura S, Fujii M, Nomura S, Suzuki M. Comparison of lumbar drainage and external ventricular drainage for clearance of subarachnoid clots after Guglielmi detachable coil embolization for aneurysmal subarachnoid hemorrhage. Clin Neurol Neurosurg. 2013 Jul;115(7):965-70. doi: 10.1016/j.clineuro.2012.10.001. Epub 2012 Oct 26. PMID 23107165
- [Background] Klimo P Jr, Kestle JR, MacDonald JD, Schmidt RH. Marked reduction of cerebral vasospasm with lumbar drainage of cerebrospinal fluid after subarachnoid hemorrhage. J Neurosurg. 2004 Feb;100(2):215-24. doi: 10.3171/jns.2004.100.2.0215. PMID 15086227